CLINICAL TRIAL: NCT07004751
Title: Determination of Etiology of Febrile Illness in Nepal (DEFINe Study)
Brief Title: Etiology of Febrile Illness in Nepal (DEFINe Study)
Acronym: DEFINe
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Patan Academy of Health Sciences (Other)
Responsible Party: Principal Investigator, Janak Koirala, Professor of Medicine and Infectious diseases, Patan Academy of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DEFINe Study
Record Dates: First submitted 2025-04-30; First posted 2025-06-04 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Febrile Illness; Fever Without Source
Keywords: Febrile Illnes

STUDY DESIGN:
Intervention Model Description: For patients without an obvious cause of fever and an inconclusive work up after standard of care evaluations, additional serological tests as a part of undifferentiated febrile illness work up will be performed including clinical evaluation; additional microbiological evaluation and laboratory testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): Standard of care evaluation of a febrile patient is done by the treating medical team which usually consists of the following set of clinical, basic laboratory, radiological and microbiological evaluations: History and Evaluation; Basic Lab Tests; Radiological Investigations; Routine Serologies; Microbiological Investigations
  Interventions: Diagnostic Test: Standard of Care (SOC)
- Study Arm (Experimental): For patients without an obvious cause of fever and an inconclusive work up after standard of care evaluations, additional serological tests as a part of undifferentiated febrile illness work up will be performed including clinical evaluation; additional microbiological evaluation and laboratory testing other than that in the standard care
  Interventions: Diagnostic Test: Additional laboratory analysis

INTERVENTIONS:
Diagnostic Test: Additional laboratory analysis — Additional lab tests will be done to establish the diagnosis of Murine typhus, Bartonellosis, Q-fever, Chikungunya, Zika, Japanese B encephalitis, West Nile virus
  Arms: Study Arm
Diagnostic Test: Standard of Care (SOC) — Standard of care evaluation of a febrile patient is done by the treating medical team as Standard of care evaluation of a febrile patient is done by the treating medical team which includes clinical, basic laboratory, radiological and microbiological evaluations
  Arms: Standard of Care

SUMMARY:
In the absence of a microbiological lab testing, majority of the cases of febrile illnesses in Nepal are diagnosed on a clinical basis alone. These cases of "undifferentiated febrile illness" are treated empirically with multiple antibiotics without an etiological diagnosis. Unnecessary use of antibiotics can increase the risk of antibiotic resistance and adds unnecessary burden of cost to the patients and their families.

This study aims to determine the etiology of infections using additional microbiological techniques in patients admitted to the hospital with acute undifferentiated febrile illness of 3 days to 21 days duration, and assess its impact on use of antimicrobial drugs. In addition to the clinical features, the etiological diagnosis will be confirmed by using additional tests including culture techniques and ELISA based serological tests for 7 additional pathogens which are currently not tested in Nepal. Patients meeting definition of undifferentiated fever of 3 days to 21 days duration will be enrolled from a major tertiary care center using predefined inclusion and exclusion criteria.This study will help to identify additional infectious diseases prevalent in Nepal, decrease unnecessary empirical use of multiple antibiotics, and improve patient outcome. Additionally, identification of new causes of febrile illness will help in prevention and control of these infectious diseases at public health level.

DETAILED DESCRIPTION:
Nepal is located between latitudes 26° and 31°N while its altitude ranges from 60m to 8848m from sea level allowing for a large variation in climate. Southern part of Nepal has tropical climate suitable for vector-borne tropical diseases whereas northern parts have more temperate and sub-arctic climate where these diseases are less common. Additionally, water-borne diseases have persisted because of a lack of sanitation and safe drinking water. Most hospitals in Nepal lack support of well equipped. microbiology laboratories for diagnosis of infectious diseases, and hence, most clinicians treat their patients empirically based on their decisions on clinical features alone . A study done in the region has shown poor predictability of clinical features alone to distinguish enteric fever from other causes of febrile illness .

Either from the lack of or limited access to confirmatory microbiological tests, majority of the cases of febrile illnesses in Nepal are diagnosed on clinical basis only. These cases of "undifferentiated fever" or "undifferentiated febrile illness" are treated empirically without etiological diagnosis. In the absence of correct diagnosis, patients receive multiple empirical antibiotics which increase the risk of antibiotic resistance and adds unnecessary burden of cost to the patients and their families. A hospital-based study of febrile patients published in 2004 revealed identifiable causes in only 37% of the patients.

The most common causes of febrile illness in Nepal at the time were enteric fever, murine typhus, scrub typhus, Leptospirosis, and bacterial infections including Streptococcus pneumoniae, Staphylococcus aureus, and Escherichia coli. Studies show a trend in increasing cases of rickettsial infections including Rickettsia typhi and Orientia tsutsugamushi.

Preliminary work done at Patan Hospital Patan Hospital is a tertiary care medical center with 450 beds that admits between 10 to 30 febrile patients per week depending on the season. Over 30% of these patients do not have localizing signs and symptoms for clinical diagnosis nor do they have a laboratory-based diagnosis. These cases are labelled as undifferentiated fever and receive empirical treatment with two or more antimicrobial agents. Previous studies done at Patan Hospital have demonstrated that Salmonella typhi and Salmonella paratyphi A were causes of undifferentiated fever of >3 days duration in 34% patients and Rickettsia typhi in 17% cases, whereas another study in 2008 found 7% cases of febrile illness has Rickettsia typhi, which is the cause of Murine typhus. These studies show an increase in cases of rickettsial infections including Riackettsia typhi and Orientia tsutsugamushi. Studies at Patan Hospital have also identified Streptococcus pneumoniae, Leptospira spp., Orientia tsutsugamushi, Hantavirus, and Coxiella burnetii as casues of febrile illnesses .

Research Gap The epidemiology of infectious disease has changed with massive within country urban migrations, increased migrant workers to India and overseas countries, change in climate, and several other reasons. Previous common causes of febrile illnesses such as malaria and enteric fever have declined over past decade whereas dengue and scrub typhus are on the rise. Meanwhile, new diseases such as COVID-19, dengue, and Scrub typhus have become commonplace [5,10,11]. Other causes of febrile illnesses, such as zoonoses (e.g. bartonellosis and Q fever), rickettsial (e.g. Q fever), and viral infections (e.g. arboviruses) remain mostly undiagnosed. This study aims to fill the gap in research by identifying additional causes and estimating burden of these infectious diseases. This will also help to reduce the unnecessary use of antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 years or older
* Documented fever (T ≥100.4F or ≥38C) of 3 days to 21 days duration
* No obvious diagnosis found on the basis of clinical, radiological, or initial routine laboratory tests*
* Admitted to the medical unit of hospital
* Signed ICF (informed consent form)

Exclusion Criteria:

* Outpatients
* Fever of less than 3 days or more than 21 days duration
* Patients being discharged from Emergency Room
* Children (younger than 16 years in age)**
* Immunocompromised patients
* Neutropenia (ANC <500 per cumm)
* Known case of HIV infection
* Admission to a hospital for 48-hours or longer within past 30 days

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2025-07-04 (Actual); Primary Completion 2026-07-10 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Estimate the etiology of fever | 0-21 days
  To estimate the proportion of additional infectious etiologies of febrile illness among patients presenting with an undifferentiated fever of 3 to 21 days duration.
Efficacy of antimicrobials | 0-21 days
  Average number of antimicrobials prescribed to participants diagnosed solely based on clinical diagnosis versus those with additional microbiological testing.

SECONDARY OUTCOMES:
appropriateness of the empiric antibiotic therapy | 0-21 days
  Percentage of participants receiving empiric antibiotic treatment with the final laboratory-confirmed diagnosis.
correlation of clinical diagnosis with laboratory diagnosis | 0-21 days
  Percentage of cases where the initial clinical diagnosis matches the laboratory-confirmed diagnosis.
Compare the Treatment outcome | 0-21 days
  Percentage of participants who gets clinical recovery by Day 21, comparing those treated based on microbiological diagnosis versus clinical diagnosis alone.

CONTACTS AND LOCATIONS:
Overall Officials: Janak Koirala, MD MPH, Principal Investigator — Patan Academy of Health Sciences
Locations (1):
- Patan Academy of Health Sciences, Lalitpur, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2025-03-01): https://cdn.clinicaltrials.gov/large-docs/51/NCT07004751/Prot_000.pdf